CLINICAL TRIAL: NCT03753906
Title: Clinical and Optical Evaluation of Self-filling Osmotic Tissue Expander in Augmenting Keratinized Tissue Around Dentulous Region
Brief Title: Evaluation of Self-filling Osmotic Tissue Expander in Augmenting Keratinized Tissue Around Dentulous Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02_D012_71909
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Soft Tissue Augmentation

STUDY DESIGN:
Intervention Model Description: All the patients were implanted with self-inflating hydrogel expander in subperiosteal positions using the pouch technique in the mandibular anterior region.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Osmed® hydrogel expander implantation (Experimental): Implantation of Osmed® hydrogel expander was done in subperiosteal positions using the pouch technique in the mandibular anterior region.
  Interventions: Device: Osmed® hydrogel expander implantation

INTERVENTIONS:
Device: Osmed® hydrogel expander implantation — Under local anaesthesia, a small vertical incision, adapted to the diameter of the Osmed® sself-inflating hydrogel expander, was made with #15 scalpel blade at the mesial line angle of the adjacent tooth which started below the gingival margin extending from the keratinized tissue above the MGJ to the non-keratinized tissue beyond the MGJ. A minimally invasive preparation of a subperiosteal pouch was performed with KPA tunnelling knife. Size of the pouch was controlled with the specific surgical template to ensure the device easily fits into the prepared pouch without tension. Expanders were secured in the correct position with a bone fixation screw, at the flat end, which does not possess an expansion capability. The wound was closed with 3-0 silk suture using simple interrupted sutures.

SUMMARY:
The present study is a human, prospective, single centre, single blind randomised controlled clinical tria conducted to explore the feasibility and efficacy of self-inflating hydrogel expander (Osmed®) to gain keratinised tissue around the dentulous area. The trial is in accordance to the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.

DETAILED DESCRIPTION:
Ten healthy individuals satisfying the inclusion and exclusion criteria were recruited for the study. A detailed, thorough medical and dental history was obtained and each patient was subjected to comprehensive clinical and radiological examination. All patients were informed about the nature of the study, surgical procedure involved, potential benefits and risks associated with the surgical procedure and a written informed consent was obtained from all patients.

All the patients were implanted with self-inflating hydrogel expander (Osmed®) in subperiosteal positions using the pouch technique in the mandibular anterior region. The clinical parameters were recorded at baseline, two weeks post expander retrieval, three months and six months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate in the study
* Patients above 18 years of age
* Systemically healthy patients
* Patients exhibiting keratinized tissue width < 2 mm
* Patients manifesting Miller's Class I or Class II recession
* Patients who demonstrate good plaque control ( PI < 10% ) and showing good compliance
* Uncompromised adjacent teeth with healthy gingival conditions

Exclusion Criteria:

* Untreated periodontal disease, caries
* Insufficient oral hygiene
* Thin biotype ( < 0.8 mm )
* Use of tobacco
* Previous radiation therapy
* Patients with known systemic diseases and conditions as uncontrolled diabetes mellitus or haemorrhagic disorders
* Pregnant and lactating women
* Non-compliant patients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11-05 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Keratinized tissue width (KTW) | 6 months
  measured from the most apical gingival margin to the mucogingival junction (MGJ), with the MGJ location determined using the visual method (Schiller's potassium iodide solution).
Keratinized tissue thickness (KTT) | 6 months
  measured at the mid-buccal aspect of the study tooth just below the marginal gingiva using an endodontic file.
Optical scanning for analysis of tissue thickness | 6 months
  alginate impressions were made at the baseline prior to expander placement, immediately after the removal of expander and 6 months post-augmentation. The prepared casts were assessed for soft tissue changes by optical scan using 3D camera (Intellidenta AG, Basel, Switzerland). The obtained digital images of the casts reflecting the different treatment time were then superimposed and matched in one common coordinate system. The buccal surfaces of the study teeth were used as a reference point for the superimposition of different images. Subsequently, a defined area of interest at each site were measured and the difference in the linear distance between the time points were calculated.

SECONDARY OUTCOMES:
Gingival recession depth (GRD) | 6 months
  measured at the mid-buccal aspect of the study tooth from the CEJ to the most apical extension of gingival margin (using UNC-15 probe)
Vestibular depth (VD) | 6 months
  measured from cemento-enamel junction (CEJ) to the deepest part of vestibular mucosa. Measurements were taken with the UNC-15 probe while exerting a firm facial pull on the lip or cheek at a 90° angle to the surface of the teeth.
Color and texture match to the surrounding tissue | 6 months
  binary ratings of "equal or not equal to surrounding native tissue" assigned upon clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Prabhuji MLV, MDS, Study Director — Krishnadevaraya College of Dental Sciences